CLINICAL TRIAL: NCT01033565
Title: Controlled-Release Melatonin (Melatonin CR)for the Treatment of Impaired Sleep Maintenance (ISM) in 4-8 Year Old Children With Autism Spectrum Disorders (ASD).
Brief Title: Melatonin CR for the Treatment of Impaired Sleep Maintenance in 4-8 Year Old Children With Autism Spectrum Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unsuccessful in recruiting appropriate subjects.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0401-09-FB
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Sleep Disorder
Keywords: Impaired sleep maintenance; Autism Spectrum Disorders; Pediatric
MeSH Terms: conditions — Sleep Wake Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Natrol (Experimental): Subjects receive Natrol (sustained release melatonin) 5mg tablet 30 minutes prior to bedtime for 10 to 14 days
  Interventions: Drug: Natrol

INTERVENTIONS:
Drug: Natrol — 5mg of sustained released melatonin. One tablet given 30 minutes prior to bedtime.
  Other Names: Sustained release melatonin

SUMMARY:
The purpose of this research is to see the effects (good and bad) of Melatonin CR on sleep in 4-8 year old children with autism spectrum disorders and sleep problems.

DETAILED DESCRIPTION:
The title of this acute, open-label pilot study is "Controlled Release Melatonin (Melatonin CR) for the treatment of impaired sleep maintenance (ISM) in 4-8 year old children with autism spectrum disorders (ASD)." Maintenance of sleep is a significant challenge in the treatment of children with neurodevelopmental disabilities including ASDs. Night awakening or early morning waking can have detrimental effects on these children's daytime behavior and the functioning of their household. Sleep problems in the ASD population are generally managed first with behavioral interventions and, when these are not successful, pharmacologic therapy. Most medications effect sleep onset and not sleep maintenance. This study investigates the effectiveness of Melatonin CR for managing ISM in 4-8 year old children with ASD. Twenty patients will be recruited from the Developmental/Behavioral Pediatrics Clinic at the Munroe Meyer Institute at the University of Nebraska Medical Center. Inclusion criteria are male and female children ages 4-8 years with a diagnosis of an ASD, including Pervasive Developmental Disorder NOS (PDD, NOS), Asperger's Syndrome, or Autistic Disorder, parent/guardian consent for participation, stable psychotropic medication treatment for at least 4 weeks, and a documented history of ISM based on parent-report, somnolog and Child Sleep Habits Questionnaire (CSHQ), and a clinician rating of ≥4 (moderately ill) on the Clinical Global Impression-Severity (CGI-S) Scale. Patients will be excluded if they have been treated with Melatonin or Melatonin CR in the past month, failed treatment with Melatonin CR, or if they have a previously un-evaluated medical condition which may be causing the ISM. Following the completion of a somnolog and standardized questionnaires, the patients will be treated for 10-14 days with melatonin CR. Somnologs will be completed during treatment, and standardized parent questionnaires, CGI-S, and adverse event collection will be repeated at the end of Melatonin CR therapy. Response will be defined as a Clinical Global Impression-Improvement (CGI-I) score of 1 or 2 (much or very much improved). These will be compared to baseline ratings. Following the completion of the study protocol, all patients will continue to be followed in the Developmental Pediatrics clinic. Data from this acute pilot trial can be used to evaluate the appropriateness of a larger study to determine optimal therapy for patients with ASD and ISM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children,
* ages 4-8 years,
* diagnosed with an ASD, including
* Pervasive Developmental Disorder NOS (PDD, NOS),
* Asperger's Syndrome, or
* Autistic Disorder, and followed in the Munroe Meyer Developmental Pediatrics Clinic. Documented impaired sleep maintenance (ISM) based on parent-report and 7 day somnolog (sleep diary).
* Clinician rating of 4 (moderately ill) or worse on CGI-S. Rating is based on the clinician's experience with evaluating and treating this patient population.
* Previous discussion during a clinic appointment about sleep difficulties, including review of sleep hygiene and basic behavioral interventions/strategies.
* Current problems of overnight awakenings recorded on the Children's Sleep Habits Questionnaire (CSHQ) despite behavioral intervention.
* Stable psychotropic medication treatment for the past 4 weeks.

Exclusion Criteria:

Treatment with Melatonin or Melatonin CR during the past month or previous failed treatment with Melatonin CR.

Presence of a previously unevaluated medical condition which may be the etiology of the nighttime awakenings. There is no contraindication for use of Melatonin CR in patients with obstructive sleep apnea.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Needelman, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center-Munroe Meyer Institute, Omaha, Nebraska, United States

REFERENCES:
- [Background] Braam W, Smits MG, Didden R, Korzilius H, Van Geijlswijk IM, Curfs LM. Exogenous melatonin for sleep problems in individuals with intellectual disability: a meta-analysis. Dev Med Child Neurol. 2009 May;51(5):340-9. doi: 10.1111/j.1469-8749.2008.03244.x. PMID 19379289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one subject was recruited who met criteria to participate.
Pre-assignment Details: One subject enrolled and finished participation.
Groups:
- Natrol: Subjects receive Natrol (sustained release melatonin) 5mg tablet 30 minutes prior to bedtime for 10 to 14 days
  Natrol : 5mg of sustained released melatonin. One tablet given 30 minutes prior to bedtime.
Period: Overall Study
Arm/Group | Natrol
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Natrol
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Improvement
Description: Assigns numerical score indicating level of improvement compared to baseline. Scale is rated from 1-7: 1= very much improved; 2= much improved; 3= minimally improved; 4= no change; 5= minimally worse; 6= much worse; 7= very much worse.
Time Frame: 2 weeks
Measure: Number; unit: units on a scale
Arm/Group | Natrol
Number analyzed (Participants) | 1
units on a scale | 2

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Natrol
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Unable to recruit a sufficient number of subjects to complete the study as designed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No